CLINICAL TRIAL: NCT05199831
Title: Preliminary Situational Analysis of a Pilot Rehabilitation Intervention Based on Physical Exercise for People Living With HIV in Ivory Coast
Brief Title: Situational Analysis of HIV-related Disability in the Context of Ivory Coast
Acronym: ViRAGE
Status: Completed | Type: Observational
Sponsor: Programme PAC-CI, Site ANRS-MIE de Côte d'Ivoire (Other)
Collaborators: Institute of Research for Development, France (Other Government); Institut de Sante Publique, d'Epidemiologie et de Developpement (Other); University of Toronto (Other); Université de Lille (Other)
Responsible Party: Sponsor
Other Study IDs: VIRAGE
Record Dates: First submitted 2021-12-14; First posted 2022-01-20 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: HIV Infections
Keywords: Aging; Disability; Functional limitations; Physical activity; Sub-Saharan Africa
MeSH Terms: conditions — HIV Infections; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants living with HIV: Clinical, functional and cognitive evaluations; questionnaires on disability, social participation, mental health and physical activity
- Controls not infected with HIV: Clinical, functional and cognitive evaluations; questionnaires on disability, social participation, mental health and physical activity

SUMMARY:
The goal of this study is to document the impairment, functional and activity limitation and disability associated with HIV infection in an African urban context.

It will combine quantitative and a qualitative methods.

The quantitative evaluation will include 300 adults living with HIV of age ≥40 years receiving antiretroviral therapy and followed at the infectious disease department (SMIT), CHU de Treichville, Abidjan, and 200 adults without HIV infection of similar age and sex (control group). This cross-sectional evaluation will combine clinical, functional and cognitive evaluations and questionnaire on disability, depression and physical activity.

The qualitative research will be based on semi-directed interviews and will examine disability perception and biographic reconstruction.

DETAILED DESCRIPTION:
Background With the scale up of antiretroviral therapy (ART), people living with HIV (PLWHIV) life expectancy has increased dramatically over the last decades and HIV has become a chronic disease. However, the long-term infection with HIV is often associated with a number of health related challenges responsible of impairments and functional limitations. To achieve the ambitious objective that most of the PLWHIV receive ART and have a good quality of life, it is therefore necessary to address the HIV-related disability.

Objectives This research aims to provide a comprehensive analysis of the frequency and nature of the impairments and functional limitation occurring in PLWHIV, and of their impact on participants lives. It will also assess the level of physical activity and the acceptability of an intervention based on physical activity.

It will adopt a multidisciplinary approach, which will combine objective and subjective measurements of disability including bio-clinical data, epidemiological data and qualitative data reflecting PLWHIV's perspective. It will also include an evaluation of the a priori acceptability of using physical exercise with PLWHIV.

Three dimensions of disability will be considered in the analysis: 1) impairment and morbidities (neurological, motor and cognitive), 2) activities (or functional) limitations, 3) social participation restrictions. The evaluation of acceptability will cover perceived relevance, adequacy, perceived efficacy and easiness of use of the intervention.

Design and methods The quantitative evaluation will include 300 PLWHIV receiving ART and followed at the infectious disease department (SMIT), CHU de Treichville, Abidjan. A control group of HV uninfected adults will also be included (n = 150). This cross-sectional evaluation will combine clinical, functional and cognitive evaluations and questionnaire on disability (WHODAS, HDQ), depression (PHQ-9) and physical exercise acceptability.

The qualitative component will include around twenty PLWHIV. Participants will be selected to reflect the diversity of the population living with HIV (regarding sex, age, family situation). The qualitative research will be based on semi-directed interviews and will examine disability perception, biographic reconstruction after the onset of impairment and the acceptability of physical exercise.

Quantitative and qualitative researches will be integrated using an explanatory sequential design. The quantitative results will be used to the qualitative research questions sampling and design. In addition, results of the two components regarding the social participation and the perception and attitude toward physical activity will be integrated.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥40 years
* HIV-1 infection (or negative HIV test within the last 12 months if control)
* Ongoing antiretroviral treatment if HIV-infected participant

Exclusion Criteria:

* Clinical symptoms suggesting an acute infection
* Any severe condition not allowing participation in the study

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants living with HIV are recruited from the Department of tropical and infectious disease at Treichville teaching hospital, Abidjan, Ivory Coast. Participants are randomly selected from the list of patients in care.
  Controls are recruited from the Blood donor centre nearby Treichville hospital. They are selected in order to match HIV-infected population distribution regarding age and sex.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2021-02-05 (Actual); Primary Completion 2022-01-10 (Actual); Study Completion 2022-08-10 (Actual)

PRIMARY OUTCOMES:
Functional capacity | Baseline
  Short Physical Performance battery (SPPB)

SECONDARY OUTCOMES:
Comorbidities: blood pressure | Baseline
  Blood pressure
Comorbidities: diabetes | Baseline
  haemoglobin glycated
Comorbidities: obesity | Baseline
  Body mass index
Neurologic outcomes CNS | Baseline
  Central nervous system abnormality
Neurologic outcomes BNPS | Baseline
  Brief Peripheral Neuropathy Score (BNPS)
Other functional scores: gate speed | Baseline
  6 minutes walk test
Other functional scores: fine motricity | Baseline
  grooved pegboard test
Other functional scores: strength | Baseline
  grip strength
Cognitive tests: color trail | Baseline
  Color trail tests 1 & 2
Cognitive tests: fluency test | Baseline
  Category words fluency test
Cognitive tests: Digit symbol substitution test (DSST) | Baseline
  Digit symbol substitution test
Cognitive tests: memory | Baseline
  Grober & Buschke test
Cognitive tests: digit span test (DST) | Baseline
  Digit span test
Disability: WHO Disability Assessment Schedule 2 (WHODAS) | Baseline
  WHODAS-2
Disability: HIV Disability Questionnaire (HDQ) | Baseline
  HDQ short form (HDQ-SF)
Disability: Instrumental Activities of Daily Life (IADL) | Baseline
  IADL assessed using the Epidemca instrument
Physical activity | Baseline
  Self reported physical activity assessed using the GPAQ instrument
Mental health: depression | Baseline
  PHQ-9
Acceptability and preference for an intervention | Baseline
  Participant preference for a possible intervention based on peer support or physical activity

CONTACTS AND LOCATIONS:
Locations (2):
- Côte d’Ivoire (2):
  - Centre National de Transfusion Sanguine, Abidjan
  - CHU Treichville, Abidjan

REFERENCES:
- [Derived] Debeaudrap P, Etoundi N, Tegbe J, Assoumou N, Dialo Z, Tanon A, Bernard C, Bonnet F, Aka H, Coffie P. The association between HIV infection, disability and lifestyle activity among middle-aged and older adults: an analytical cross-sectional study in Ivory Coast (the VIRAGE study). BMC Public Health. 2024 Jun 8;24(1):1549. doi: 10.1186/s12889-024-19020-9. PMID 38851706